CLINICAL TRIAL: NCT05405621
Title: A Phase 1, Multi-Center, Open-Label Study to Assess Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of BAT8009 in Patients With Advanced Solid Tumours
Brief Title: Assess Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of BAT8009
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-8009-001-CR
Record Dates: First submitted 2022-05-30; First posted 2022-06-06 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Locally Advanced/Metastatic Solid Tumours
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Experimental): Experimental: BAT8009 for Injection 0.6 mg/kg (frequency: Q3W)
  Interventions: Drug: BAT8009 for Injection
- Cohort 2 (Experimental): Drug: BAT8009 for Injection 1.2 mg/kg (frequency: Q3W)
  Interventions: Drug: BAT8009 for Injection
- Cohort 3 (Experimental): Drug: BAT8009 for Injection 2.4 mg/kg (frequency: Q3W)
  Interventions: Drug: BAT8009 for Injection
- Cohort 4 (Experimental): Drug: BAT8009 for Injection 3.6mg/kg (frequency: Q3W)
  Interventions: Drug: BAT8009 for Injection
- Cohort 5 (Experimental): Drug: BAT8009 for Injection 4.8mg/kg (frequency: Q3W)
  Interventions: Drug: BAT8009 for Injection
- Cohort6 (Experimental): Drug: BAT8009 for Injection 6.0mg/kg (frequency: Q3W)
  Interventions: Drug: BAT8009 for Injection
- Cohort 7 (Experimental): Drug: BAT8009 for Injection 7.2mg/kg (frequency: Q3W)
  Interventions: Drug: BAT8009 for Injection
- Cohort 8 (Experimental): Drug: BAT8009 for Injection 8.4mg/kg (frequency: Q3W)
  Interventions: Drug: BAT8009 for Injection

INTERVENTIONS:
Drug: BAT8009 for Injection — BAT8009 will be administered as a 90-minute (± 5min) IV infusion on Day 1 of Cycle 1. If there is no infusion related reaction after initial dose, the next dose of BAT8009 will be infused intravenously into each patient for approximately 30~120 minutes.
  Other Names: Recombinant Humanized Anti-B7H3 Monoclonal Antibody-Exatecan Conjugate

SUMMARY:
Primary objectives:

* To evaluate the safety and tolerability of BAT8009 in patients with advanced solid tumours.
* To determine the maximum tolerated dose (MTD) and recommended dose for Phase 2 (RP2D).

DETAILED DESCRIPTION:
This is a first-in-human (FIH), multicentre, open-label, Phase 1 dose escalation and dose expansion study of BAT8009 (a B7H3-targeting antibody-drug conjugate) in patients with advanced solid tumours.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give voluntary informed consent and understand the study and are willing to follow and complete all the study required procedures.
2. Aged ≥ 18 years and ≤ 75 years.
3. Life expectancy ≥ 3 months.
4. ECOG performance status ≤ 1.
5. Histologically/cytologically confirmed, locally advanced unresectable or metastatic solid tumours that are refractory to standard therapy.
6. Has measurable or evaluable disease per RECIST v1.1.
7. Adequate haematological, liver, kidney, cardiac and coagulation function.
8. Is willing to provide pre-existing diagnostic or resected tumour samples (if available).
9. Female patients must: Be of non-child-bearing potential; Male patients must: be willing not to donate sperm.
10. Must agree to adhere to the current state and national advice regarding minimising exposure to COVID-19 from the first Screening visit until the end of study (28-day Safety Follow-up Visit).

Exclusion Criteria:

1. Females who are pregnant or nursing.
2. Receiving concurrent anticancer therapy or investigational therapy.
3. Persisting AEs that are > Grade 1 from prior antitumour treatment as per CTCAE v5.0.
4. Patients with primacy central nervous system (CNS) malignancy, symptomatic CNS metastases, meningeal metastases or leptomeningeal disease are not allowed.
5. Had major surgery within 28 days of the Screening visit.
6. History of autologous transplantation ≤ 3 months.
7. History of severe infection deemed clinically significant by the PI or designee within 4 weeks.
8. History of human immunodeficiency virus (HIV) infection.
9. Active hepatitis B or C.
10. History of a Grade 3 or Grade 4 allergic reaction to treatment with other antibodies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | A minimum of 21 days after first dose of BAT8009
  A DLT is defined as a toxicity occurring during the DLT observation period

SECONDARY OUTCOMES:
Cmax (Maximum serum concentration) | 126 days after first dosing
  Maximum observed plasma or serum concentration
Immunogenicity | 126 days after first dosing
  Presence of ADAs / neutralizing antibodies (NAbs).
AUC0-inf after Cycle 1 administration and AUC0- λ after Cycle 6 administration | 126 days after first dosing
  area under the serum concentration versus time curve from time zero to infinity and to time λ

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD